CLINICAL TRIAL: NCT02256189
Title: The Effect of Sitagliptin on Glucagon Counterregulation and Incretin Hormones During Mild Hypoglycemia in Elderly Patients With Metformin-treated Type 2 Diabetes
Brief Title: Sitagliptin and Glucagon Counterregulation
Acronym: SITACLAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 300A
Record Dates: First submitted 2014-09-29; First posted 2014-10-03 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin first, then placebo (Other): Sitagliptin treatment for four weeks, then washout for four weeks, then placebo for four weeks
  Interventions: Drug: Sitagliptin
- Placebo first, then sitagliptin (Other): Placebo for four weeks, then washout for four weeks, then sitagliptin for four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg daily
  Arms: Sitagliptin first, then placebo
Drug: Placebo — Placebo one tablet daily
  Arms: Placebo first, then sitagliptin

SUMMARY:
To evaluate the effect of DPP-4 inhibition on glucagon counter-regulatory mechanisms at moderate hypoglycemia in metformin-treated subjects with T2DM

DETAILED DESCRIPTION:
The glucagon response to mild (3.0 mmol/l) hypoglycemia with and without DPP-4 inhibition by sitagliptin will be evaluated in elderly subjects with metformin treated type 2 diabetes to explore whether DPP-4 inhibition affects glucagon counter-regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent has been given.
2. Patients with metformin treated T2DM (metformin dose >0,5 g/day and stable during the preceding 3 months)
3. Age >65 years.
4. HbA1c 6.0-8.5% (43-67 mmol/mol; inclusive) at visit 1.
5. Ability to complete the study

Exclusion Criteria:

1. A history of any secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly.
2. Type 2 diabetes, positive GAD antibodies
3. eGFR <60 ml/min
4. Acute infections which may affect blood glucose control within 4 weeks prior to visit 1
5. Any history of recent (<2 weeks) recurrent or severe hypoglycemic episodes.
6. Liver disease such as cirrhosis or chronic active hepatitis
7. History of coronary heart disease or heart failure class III or IV
8. Donation of one unit (500 ml) or more of blood, significant blood loss equaling to at least one unit of blood within the past 2 weeks or a blood transfusion within the past 8 weeks.
9. Treatment with growth hormone of chronic oral or parenteral corticosteroid treatment (> 7 consecutive days of treatment) within 8 weeks prior to visit 1.
10. Use of other investigational drugs at visit 1 or within 30 days of visit 1, unsuitable for the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Skane University Hospital Malmö, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin First, Then Placebo: Sitagliptin first for four weeks, then washout for four weeks, then placebo for four weeks
- Placebo First, Then Sitagliptin: Placebo first for four weeks, then washout for four weeks, then placebo for four weeks
Period: Overall Study
Arm/Group | Sitagliptin First, Then Placebo | Placebo First, Then Sitagliptin
Started | 15 | 13
Completed | 15 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin First, Then Placebo: Hypoglycemia clamp with sitagliptin
  Sitagliptin: Treatment with sitagliptin 100mg QD for four weeks followed by hyperinsulinemic hypoglycemic clamp
- Placebo First, Then Stagliptin: Hypoglycemia clamp with placebo
  Placebo: Treatment with placebo QD for four weeks followed by hyperinsulinemic hypoglycemic clamp
- Total: Total of all reporting groups
Arm/Group | Sitagliptin First, Then Placebo | Placebo First, Then Stagliptin | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 75.0 (5.9) | 71.9 (5.7) | 73.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 15 | 13 | 28
Fasting glucagon [Mean (Standard Deviation); unit: pmol/l] | 29.5 (9.7) | 30.0 (12.2) | 29.8 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Glucagon Counterregulation to Hypoglycemia
Description: Change in plasma glucagon to insulin-induced hypoglycemia after four weeks of treatment with sitagliptin and placebo
Time Frame: Four weeks treatment
Measure: Mean (Standard Error); unit: pmol/l
Groups:
- Sitagliptin: Hypoglycemia clamp with sitagliptin
  Sitagliptin: Treatment with sitagliptin 100mg QD for four weeks followed by hyperinsulinemic hypoglycemic clamp
- Placebo: Hypoglycemia clamp with placebo
  Placebo: Treatment with placebo QD for four weeks followed by hyperinsulinemic hypoglycemic clamp
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 28 | 28
pmol/l | 16.0 (2.9) | 16.5 (2.8)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Placebo First, Then Stagliptin: Placebo first for four weeks, then washout for four weeks, then sitalgiptin for four weeks
- Sitagliptin: Sitagliptin 100mg Daily for four weeks, either before or after a 4 week placebo period
- Placebo: Placebo Daily for four weeks, efter before or after a 4 week sitagliptin period
Arm/Group | Sitagliptin First, Then Placebo | Placebo First, Then Stagliptin | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02256189/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02256189/SAP_001.pdf